CLINICAL TRIAL: NCT01800045
Title: A Randomized, Double Blind Study Comparing Pitolisant (BF2.649) to Placebo in Two Parallel Groups on the Weekly Frequency of Cataplexy Attacks and Excessive Daytime Sleepiness in Narcoleptic Patients With Cataplexy.
Brief Title: Pitolisant to Assess Weekly Frequency of Cataplexy Attacks and EDS in Narcoleptic Patients (HARMONY CTP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P11-05 / Pitolisant; 2012-003076-39 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-27 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2015-07

CONDITIONS: Narcolepsy With Cataplexy; Excessive Daytime Sleepiness
Keywords: Narcolepsy; Cataplexy; Sleep disorder; Excessive daytime sleepiness
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence; Cataplexy; Sleep Wake Disorders | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitolisant (Experimental): Pitolisant at 5, 10, 20 or 40mg
  Interventions: Drug: Pitolisant
- Placebo (Placebo Comparator): Capsules of placebo containing lactose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitolisant — 1 capsule in the morning before breakfast
  Other Names: BF2.649
  Arms: Pitolisant
Drug: Placebo — 1 capsule in the morning before breakfast
  Other Names: Capsules of placebo containing lactose
  Arms: Placebo

SUMMARY:
Double blind, randomized, parallel groups study of Pitolisant versus placebo, in narcoleptic patients experiencing EDS, and cataplexy (minimum of 3 complete or partial cataplexy attacks per week).

The patients will be treated during 7 weeks with Pitolisant or placebo.

DETAILED DESCRIPTION:
The treatment period (7 weeks double blind) will aim at demonstrating the efficacy of Pitolisant on the number of cataplexy attacks and the Excessive Daytime Sleepiness by verifying whether the results of Pitolisant are superior to those of placebo.

The safety will also be assessed.

ELIGIBILITY:
Main Inclusion Criteria:

* Narcoleptic with cataplexy : at least 3 weekly cataplexy attacks
* ESS > or = 12
* ICF signed and dated

Main Exclusion Criteria:

* Other conditions that could generate EDS
* Psychological and neurological disorders
* Acute or chronic severe disease
* Treatment by prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Measure of anticataplectic efficacy | At week 7
  Measure of anticataplectic efficacy assessed by the change in the average number of cataplexy attacks per week.

SECONDARY OUTCOMES:
Excessive Daytime Sleepiness assessment | At week 7
  Excessive Daytime Sleepiness assessment by evaluation of ESS score, and other questionnaires.
Safety assessment | 11 weeks
  Safety assessment thanks to AE recording, vitals signs assessment, ECG...

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne De Paillette, Dr, Study Director — Bioprojet
Locations (1):
- State Health Center, Budapest, Hungary

REFERENCES:
- [Derived] Meskill GJ, Davis CW, Zarycranski D, Doliba M, Schwartz JC, Dayno JM. Clinical Impact of Pitolisant on Excessive Daytime Sleepiness and Cataplexy in Adults With Narcolepsy: An Analysis of Randomized Placebo-Controlled Trials. CNS Drugs. 2022 Jan;36(1):61-69. doi: 10.1007/s40263-021-00886-x. Epub 2021 Dec 21. PMID 34935103
- [Derived] Watson NF, Davis CW, Zarycranski D, Vaughn B, Dayno JM, Dauvilliers Y, Schwartz JC. Time to Onset of Response to Pitolisant for the Treatment of Excessive Daytime Sleepiness and Cataplexy in Patients With Narcolepsy: An Analysis of Randomized, Placebo-Controlled Trials. CNS Drugs. 2021 Dec;35(12):1303-1315. doi: 10.1007/s40263-021-00866-1. Epub 2021 Nov 25. PMID 34822113
- [Derived] Szakacs Z, Dauvilliers Y, Mikhaylov V, Poverennova I, Krylov S, Jankovic S, Sonka K, Lehert P, Lecomte I, Lecomte JM, Schwartz JC; HARMONY-CTP study group. Safety and efficacy of pitolisant on cataplexy in patients with narcolepsy: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2017 Mar;16(3):200-207. doi: 10.1016/S1474-4422(16)30333-7. Epub 2017 Jan 25. PMID 28129985